CLINICAL TRIAL: NCT02861638
Title: Effects of Action Observation Therapy in Patients Recovering From Total Hip Arthroplasty: A Prospective Clinical Trial
Brief Title: Action Observation in Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Jorge Hugo Villafañe, PhD, Researcher, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hip Replacement
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Total Hip Replacement
Keywords: Total hip replacement; Action observation treatment; Rehabilitation; Arthroplasty
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Video of the exercises and conventional physiotherapy. 30 minutes twice a day, 5 days a week for 2 weeks.
  Interventions: Device: Experimental group; Device: Conventional physiotherapy
- Control group (Active Comparator): Video of nature scenes and conventional physiotherapy. 30 minutes twice a day, 5 days a week for 2 weeks.
  Interventions: Device: Control group; Device: Conventional physiotherapy

INTERVENTIONS:
Device: Experimental group — Video of the exercises
  Arms: Experimental group
Device: Control group — video of nature scenes
  Arms: Control group
Device: Conventional physiotherapy — Mobilization, exercises and transfer practice.

SUMMARY:
Postoperative rehabilitation is required for a successful outcome following total hip arthroplasty. Traditionally rehabilitative programs aim to increase range of motion, to strengthen quadriceps, to restore normal gait, and to recover independence in activities of daily living. In the last decade action observation treatment, in addition to conventional physiotherapy has been proposed as a treatment method in rehabilitative medicine. There is growing evidence of the applicability of action observation training in rehabilitative medicine, indeed it has been applied in the rehabilitation of stroke of Parkinson disease of cerebral palsy and of aphasia.

Nevertheless those are small studies and one of them included a mixed population of hip and knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip replacement.

Exclusion Criteria:

* bilateral hip replacement
* previous total hip replacement.
* pre-existing motor impairment (i.e. hemiparesis, poliomyelitis, lumbar sciatica);

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change of Pain intensity | Baseline and immediately post-intervention
  Visual Analogue Scale (VAS)
Change of Range Of Motion (ROM) | Baseline and immediately post-intervention
  Active and passive range of motion of hip

SECONDARY OUTCOMES:
Barthel index | Baseline and immediately post-intervention
  Barthel Index of Activities of Daily Living
Short Form-36 motor | Baseline and immediately post-intervention
  The Medical Outcome Study 36-Item Short Form Health Survey (SF-36) is a widely used method to evaluate health-related quality of life
Tinetti scale | Baseline and immediately post-intervention
  Balance
Lequesne index | Baseline and immediately post-intervention
  The Lequesne Index is a 10-question survey given to patients with osteoarthritis of the knee

CONTACTS AND LOCATIONS:
Overall Officials: JORGE H VILLAFAÑE, PhD, Principal Investigator — IRCCS Don Gnocchi Foundation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Villafane JH, Pirali C, Isgro M, Vanti C, Buraschi R, Negrini S. Effects of Action Observation Therapy in Patients Recovering From Total Hip Arthroplasty Arthroplasty: A Prospective Clinical Trial. J Chiropr Med. 2016 Dec;15(4):229-234. doi: 10.1016/j.jcm.2016.08.011. Epub 2016 Oct 5. PMID 27857630
- See also: Exercises video — https://youtu.be/UJx5u2LmNok